CLINICAL TRIAL: NCT05690620
Title: The Effect of Laughter Yoga on Happiness and Stress in Nursing Cells Which Have Been Used for the First Time in Clinical Practice
Brief Title: Laughter Yoga for Nursing Students Going Into Clinical Practice for the First Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Betül Bal
Record Dates: First submitted 2023-01-06; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Happiness; Laughter Yoga; Nursing Student; Stress; Clinical Practice
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga (Experimental): In a systematic review study, it was determined that it was appropriate to practice laughter yoga for at least 4 weeks. Therefore, the laughter yoga program; It was planned as a face-to-face group session, for four (4) weeks, twice a week, for a total of eight (8) sessions and 20-25 minutes.
  Interventions: Behavioral: laughter yoga
- Control (Active Comparator): No intervention will be applied to the students in the control group. Students will be followed for four weeks. Before the study, data collection tools will be applied to the students. Again, after the study starts and the study ends, all other data collection tools except the "Student Information Form" will be applied.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: laughter yoga — Therefore, the laughter yoga program; It was planned as a face-to-face group session, for four (4) weeks, twice a week, for a total of eight (8) sessions and 20-25 minutes.
  Arms: Laughter Yoga
Other: Control — The students in the control group did not receive any intervention. Nursing students were followed for four weeks. Before the study, data collection tools were applied to the students. Again, after the start of the study and the end of the study, all other data collection tools except the "Student Information Form" were applied.
  Arms: Control

SUMMARY:
Clinical practice is an unseparated part of nursing curricula and crucial for students to learn professional skills and gain professional identity. Besides, the clinical practices have an important role in the development of professional identity, are also emotionally challenging and stressful. All these experiences can negatively affect the happiness of nursing students. The unhappiness and stress affect nursing students negatively in terms of their physical and mental health, and lead to decreased performance, increased risk of error, and decreased quality of nursing care. Additionally, nursing students' perspectives on the profession might be negatively affected. Therefore, increased the level of happiness and reduced stress level in nursing students is important in the clinical learning environment.

Study authors could not find any studies which examining the effect of laughter yoga on the level of happiness and stress in nursing students who experienced clinical practice for the first time. Therefore, this project aimed to examine the effect of laughter yoga on the happiness and stress levels of nursing students. Study population composed of 61 students studying in the nursing department of a university located in the Central Anatolia Region. Students included in the study will be randomized into intervention and control groups according to a simple randomization rule. A total of 8 sessions of laughter yoga will be applied to the intervention group by the primary researcher for 4 weeks. Personal Information Form, Happiness Scale and Perceived Stress Scale for Nursing Students will be used as data collection tools in the research. Data collection tools will be applied in the form of pre-test and post-test. within the scope of this project, increased students' happiness and decreased stress levels were expected.

DETAILED DESCRIPTION:
Clinical practice in nursing education; It is a process that gives the opportunity to transfer knowledge into practice, gains experience and also enables the transition from student to professionalism . This process; Nursing students face many difficulties and negatively affect the sense of happiness, which is one of the basic human needs. Increasing happiness in nursing students, on the other hand, helps to positively affect quality nursing care by supporting physical and mental health, which is important for patient care. Also happiness; it reduces nursing care errors by increasing resilience, life satisfaction and performance. Happiness is expressed as a cognitive assessment of life satisfaction based on experience. However, current evidence shows that nursing students have low levels of happiness. Happiness is very important in the training and development of nursing students as future nurses; because people are more willing to help others when they are happy. When nursing students live a happy life and have personal qualities that will create happiness in others, they may be interested in caring for their patients and ensuring their happiness. However, some studies report that nursing students may experience psychological problems such as increased stress levels as well as unhappiness due to the intense curriculum and difficulties in clinical practice.

Clinical practice, which prepares students for professional nursing roles and aims to improve their clinical decision-making skills, can cause stress in students. Since the 1970s, many researchers have investigated clinical practice-related stress in nursing students and identified it as one of the major problems worldwide. Stress is a situation that challenges or exceeds the individual's coping methods of internal and external demands or both. Therefore, going into clinical practice for the first time is considered one of the important factors that cause stress in nursing students. Current evidence shows that nursing students experience moderate to high levels of stress related to clinical practice. Factors causing stress; fear of uncertainty, engaging in various clinical activities, dealing with patients, lack of knowledge and skills, fear of failure, clinical inadequacy, fear of making mistakes, lack of control associated with patients, and the experience of witnessing death. In addition, situations such as lack of communication with interdisciplinary team members, avoidance of peers and clinicians are among the factors that cause stress. Any of these factors can negatively affect the education process of the nursing student and reduce their academic performance. In addition, unhappiness and increased stress levels can negatively affect clinical learning outcomes and clinical competence. When the literature was examined, it was seen that the studies focused on reducing the stress of the students who went into clinical practice. In these studies, it was emphasized that nursing interventions such as mindfulness and peer support were effective in reducing stress.

Laughter yoga, which is one of the stress-reducing methods based on laughter; It is a type of exercise that combines unconditional laughter and breathing techniques. In this exercise method; one begins to laugh without first being a humor, a joke, or a funny incident. Natural and imitated laughter cannot be distinguished by the brain; It is known to have similar effects on the body, such as decreasing muscle tone and increasing muscle relaxation by stimulating the parasympathetic system. Laughter yoga; It helps to improve interpersonal relationships by reducing negative emotions such as tension, anxiety, hatred and anger, and relieving stress and depression in individuals. Stated that laughter yoga positively affects general health, improves sleep disorder symptoms, decreases anxiety and depression levels, and improves social functions. Confirming this view, some studies have also found that laughter yoga reduces depression symptoms, anxiety and stress levels. In addition, self-confidence, happiness, energy, positively affects memory, creative thinking and problem-solving ability; it increases interpersonal relationships, social interaction, cooperation, group identity and solidarity. In addition, laughter yoga is a very effective and practical method as it is low cost and can be performed easily regardless of time. In the light of this information, it is seen that laughter yoga is practiced in samples of patients diagnosed with diabetes, end-stage renal failure and cancer, the elderly, postpartum and menopausal women, students and individuals in the general society.

Laughter yoga sessions with nursing students have been shown to have positive effects on stress, happiness, general health and anxiety levels. However, no study has been found in the literature examining the effect of laughter yoga on happiness and stress levels in nursing students who are practicing for the first time. Laughter yoga may have a positive effect on the happiness and stress levels of nursing students who are in clinical practice for the first time. Thus, it is thought that the laughter yoga that will be applied within the scope of the project will increase the happiness level and reduce the stress level of the nursing students who will go into clinical practice for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* First time clinical practice

Exclusion Criteria:

* Inactive student registration
* Diagnosed with cardiovascular disease such as hypertension and arrhythmia
* Having had an abdominal hernia, an abdominal operation (within 3 months),
* Diagnosed with glaucoma and epilepsy
* Being on medication for psychiatric reasons
* Have experience of laughter yoga
* Using other relaxation techniques with a similar effect at the time of the study

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Happiness Level | 4 weeks
  This form will be used to measure the degree of happiness in nursing students. In the research, it will be applied twice in total, before the laughter yoga is applied and after the laughter yoga is finished. The total score to be taken from the scale varies between 6 and 30, and as the score increases, the level of happiness also increases.

SECONDARY OUTCOMES:
Change in Perceived Stress Level for Nursing Students | 4 weeks
  This form will be used to measure the level of stress in nursing students. In the research, it will be applied twice in total, before the laughter yoga is applied and after the laughter yoga is finished. The scale total score ranges from 0 to 116. A high score indicates a high level of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Betül, Yozgat, Turkey (Türkiye)